CLINICAL TRIAL: NCT03907098
Title: A Phase II Study of Endostar in Combination With Chemotherapy in HER-2 Negative Advanced Breast Cancer
Brief Title: Endostar in Combination With Chemotherapy in HER-2 Negative Advanced Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Xiaojia Wang(xj wang), Director, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZJCHBC008
Record Dates: First submitted 2019-03-29; First posted 2019-04-08 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer
Keywords: breast cancer; endostar
MeSH Terms: conditions — Breast Neoplasms | interventions — endostar protein; Endostatins; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- endostar + chemotherapy (Experimental): Endostar 15 mg per square of BSA, continuous intravenous infusion 24 hours a day, continuous administration for 7 days, every three weeks.
  Chemotherapy regimens are selected by physicians based on regular clinical decision.
  Interventions: Drug: Endostar; Drug: Chemotherapy

INTERVENTIONS:
Drug: Endostar — an anti-angiogenesis drug
  Other Names: Recombinant human endostatin
Drug: Chemotherapy — Physician's choice

SUMMARY:
This research study is studying endostar in combination with chemotherapy as a possible treatment for HER-2 negative advanced breast cancer.

DETAILED DESCRIPTION:
This is a multi-center phase II open label single-arm study to assess the safety and efficacy of endostar in combination with chemotherapy for patients with locoregionally recurrent or metastatic HER-2 negative breast cancer.

Endostar is an anti-angiogenesis drug. It is prepared by adding 9 amino acids to the N-terminal of the peptide chain on the basis of endostatin. Studies have shown that there may be a synergistic effect between endostar and chemotherapeutic agents.

ELIGIBILITY:
Inclusion Criteria:

* locoregionally Recurrent or metastatic breast cancer confirmed by histology.
* HER-2 Negative Breast Cancer.
* At least one measurable lesion according to RECIST 1.1..
* Chemotherapy for recurrent and metastatic lesions should be discontinued for more than 2 weeks.
* 18-70 years old.
* ECOG PS 0～1.
* Participants must have normal organ and marrow function as defined below: ANC ≥ 1.5×109/L,PLT ≥ 75×109/L,Hb ≥ 100 g/L;TBIL≤1.0ULN；ALT and AST≤3×ULN（ALT and AST≤5×ULN if liver metastasis）;BUN and Cr≤1.5×ULN and CCr≥50 mL/min.
* life expectancy is not less than 12 weeks.
* Signed informed consent.

Exclusion Criteria:

* Uncontrolled central nervous system metastasis.
* Not recovered to 0-1 degree (CTC AE 4.0) from toxic reactions of previous treatments..
* History of allergy to biological agents in the past.
* Important organ dysfunction and severe heart disease, including congestive heart failure, uncontrollable arrhythmia, angina, valvular disease, myocardial infarction, and refractory hypertension.
* Pregnant or lactating women..
* The patient had a history of other malignant tumors, except for the cured skin basal cell carcinoma and cervical cancer.
* The risk of uncontrolled infection, thrombosis and bleeding exists.
* A history of immunodeficiency, including HIV positive, HCV, active hepatitis B, or other acquired, congenital immunodeficiency disorders, or organ transplantation, is known.
* Researchers consider it inappropriate to carry out the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-06-30 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | up to approximately 100 months
  From enrollment to disease progression or death due to any cause

SECONDARY OUTCOMES:
Overall Survival (OS) | up to approximately 100 months
  From enrollment to death due to any cause
Objective Response Rate (ORR） | up to approximately 100 months
  Ratio of CR and PR in all subjects
Clinical Benefit Rate (CBR) | up to approximately 100 months
  Ratio of CR,PR and SD more than or equal to 24 weeks
Adverse events (AEs) | from enrollment to 30 days after the last dose administration
  Described in terms of CTC AE 4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided